CLINICAL TRIAL: NCT01739959
Title: Raised Serum Lactate as a Marker of Necrotizing Fasciitis; a Consecutive Prospective Review.
Brief Title: Exploratory Study of Raised Serum Lactate as a Marker of Necrotizing Fasciitis
Status: Completed | Type: Observational
Sponsor: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, George Murphy, Principal Investigator, National Health Service, United Kingdom
Other Study IDs: WPH/NF/2000-2010
Record Dates: First submitted 2012-11-26; First posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Fasciitis, Necrotizing
Keywords: Necrotizing fasciitis; Fournier's gangrene; Cellulitis; Serum Lactate
MeSH Terms: conditions — Fasciitis, Necrotizing; Fournier Gangrene; Cellulitis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Necrotizing fasciitis proven: Histological evidence of necrotizing fasciitis at initial surgical debridement
- Not necrotizing fasciitis: A composite of those with no histological tissue necrosis at initial surgical debridement, and those clinically judged not to be a necrotizing infection who therefore did not undergo surgery.

SUMMARY:
The investigators examined the hypothesis that serum lactate is raised in early necrotizing fasciitis to a much greater extent than in other differential diagnoses, such as severe cellulitis, and therefore provides a diagnostic indicator.

DETAILED DESCRIPTION:
A prospective comparison of serum lactate levels at referral to the Plastic Surgery team to the 'gold standard' test of histology at initial surgical debridement, looking at 53 consecutive patients referred with suspected necrotizing fasciitis to a single surgeon at one institution between 2000 and 2010.

ELIGIBILITY:
Inclusion Criteria:

* Referral to one consultant (Mr A Armstrong) at one institution (Wexham Park Hospital) with a suspected diagnosis of necrotizing fasciitis between September 2000 and September 2010

Exclusion Criteria:

* Nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients referred to a single surgeon at one institution over 10 years (September 2000 - September 2010) with a suspected diagnosis of necrotizing fasciitis. Patients were followed for the duration of their hospital stay.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2000-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Serum lactate level | At referral to the Plastic Surgery Team
  Serum lactate level at initial referral to the plastic surgery team, as measured by arterial blood gas analysis (calibrated point-of-care testing). Levels compared between the group with confirmed histological necrosis at initial surgical debridement, versus those with no evidence of necrosis (a composite of those who did not undergo surgery as they were judged not to have necrotizing fasciitis, and those who did undergo surgery, but whose histology did not show tissue necrosis).

CONTACTS AND LOCATIONS:
Overall Officials: George Murphy, MRCS, Principal Investigator — Wexham Park Hospital
Locations (1):
- Wexham Park Hospital, Slough, London, United Kingdom